CLINICAL TRIAL: NCT06072326
Title: Individual and Combined Endothelin Receptor and SGLT2 Antagonism in Adults With Type 1 Diabetes Mellitus and Chronic Kidney Disease: a Phase 2, Multicenter, Open-label Randomized Cross-over Trial
Brief Title: dApagliflozin SC0062 and Prevention of Renal Injury; a Randomized Evaluation
Acronym: ASPIRE-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17042; 2023-504404-28-00 (EU CTIS Number)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes Mellitus With Diabetic Nephropathy
Keywords: Diabetic kidney disease; sodium glucose co-transporter 2 inhibitors; endothelin receptor antagonists; Type 1 Diabetes; combination therapy
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 1 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label randomized cross-over trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment order 1 (Experimental): Subjects will start with 4 weeks of SC0062 in treatment period 1. In period 2 subjects will receive dapagliflozin. In period 3 subjects will receive a combination of SC0062 and dapagliflozin. Between treatment periods there is a 4-week wash-out.
  Interventions: Drug: Dapagliflozin (Forxiga®); Drug: SC0062 strength 10mg; Drug: SC0062 and dapagliflozin
- Treatment order 2 (Experimental): Subjects will start with 4 weeks of SC0062 in treatment period 1. In period 2 subjects will receive a combination of SC0062 and dapagliflozin. In period 3 subjects will receive dapagliflozin. Between treatment periods there is a 4-week wash-out.
  Interventions: Drug: Dapagliflozin (Forxiga®); Drug: SC0062 strength 10mg; Drug: SC0062 and dapagliflozin
- Treatment order 3 (Experimental): Subjects will start with 4 weeks of dapagliflozin in treatment period 1. In period 2 subjects will receive a combination of SC0062 and dapagliflozin. In period 3 subjects will receive SC0062. Between treatment periods there is a 4-week wash-out.
  Interventions: Drug: Dapagliflozin (Forxiga®); Drug: SC0062 strength 10mg; Drug: SC0062 and dapagliflozin
- Treatment order 4 (Experimental): Subjects will start with 4 weeks of dapagliflozin in treatment period 1. In period 2 subjects will receive SC0062. In period 3 subjects will receive a combination of SC0062 and dapagliflozin. Between treatment periods there is a 4-week wash-out.
  Interventions: Drug: Dapagliflozin (Forxiga®); Drug: SC0062 strength 10mg; Drug: SC0062 and dapagliflozin
- Treatment order 5 (Experimental): Subjects will start with 4 weeks of a combination of SC0062 and dapagliflozin in period 1. In period 2 subjects will receive SC0062. In period 3 subjects will receive dapagliflozin. Between treatment periods there is a 4-week wash-out.
  Interventions: Drug: Dapagliflozin (Forxiga®); Drug: SC0062 strength 10mg; Drug: SC0062 and dapagliflozin
- Treatment order 6 (Experimental): Subjects will start with 4 weeks of a combination of SC0062 and dapagliflozin in period 1. In period 2 subjects will receive dapagliflozin. In period 3 subjects will receive SC0062. Between treatment periods there is a 4-week wash-out.
  Interventions: Drug: Dapagliflozin (Forxiga®); Drug: SC0062 strength 10mg; Drug: SC0062 and dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin (Forxiga®) — 5 mg/day as a tablet
Drug: SC0062 strength 10mg — 20 mg/day, twice daily, capsule
Drug: SC0062 and dapagliflozin — 20 mg/day SC0062 10 mg twice daily as a capsule in combination with 5 mg/day dapagliflozin 5 mg as a tablet

SUMMARY:
The aim of this study is to test the hypothesis that dapagliflozin (SGLT2 inhibitor) and SC0062 (ERA) combination therapy augments nephroprotection and mitigates fluid retention and ketogenesis in people with T1D through complementary and synergistic mechanisms of actions.

DETAILED DESCRIPTION:
A phase 2, multicenter, randomized, open-label, cross-over trial will be conducted in male or female individuals (N=36) diagnosed with type 1 diabetes at least 6 months prior to informed consent aged between 18 and 65 years, Body Mass Index (BMI) ≥ 21 kg/m2, urinary albumin: creatinine ratio ≥ 50 mg/g and < 3000 mg/g, eGFR > 30 and <90 mL/min/1.73 m2 and HbA1c > 6.5 and <10.5%. Patients have to be on stable RAAS inhibition for at least 4 weeks prior to screening.

The study will consist of a screening visit, a 4-week run-in phase. After the run-in phase, the participant will be randomized to treatment of SC0062, dapagliflozin, or their combination in random order. The duration of each treatment period is 4 weeks with study visits scheduled at 2 and 4 weeks in each treatment period. At the end of each treatment period patients proceed to a 4 weeks wash-out phase to study off drug effects. The total duration of the study for each participant after randomization is thus 24 weeks

Interventions SC0062 10mg twice daily (20mg/day); dapagliflozin 5mg once daily; combination of SC0062 10mg twice daily and dapagliflozin 5mg once daily.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign informed consent
* Male or female individuals diagnosed with type 1 diabetes at least 6 months prior to informed consent
* WOCBP must have a negative pregnancy test at screening and must not be lactating.
* Male individuals must use highly effective method of contraception for the duration of the study (from the time they sign consent) and for 4 weeks after the last dose of study medication, or be able to provide proof of vasectomy.
* Female individuals must use highly effective method of contraception for the duration of the study (from the time they sign consent) and for 4 weeks after the last dose of study medication, provide proof of hysterectomy or sterilization, or be deemed menopausal based on a FSH-test.
* Age ≥18 and <65years, at the time of signing consent.
* Body Mass Index ≥ 21 kg/m2
* Urinary albumin:creatinine ratio ≥ 50 mg/g and <3000 mg/g
* eGFR ≥30 and <90 ml/min/1.73m2
* Stable RAAS inhibition medication for at least 4 weeks prior to screening
* HbA1c ≥6.5 and <10.5%.
* Based on the Investigator's judgment participant must have a good understanding of his/her disease and how to manage it, and be willing and capable of performing the following study assessments (assessed before randomization):

  * patient-led management and adjustment of insulin therapy
  * reliable approach to insulin dose adjustment for meals, such as carbohydrate counting
  * reliable and regular home-based blood glucose monitoring
  * established "sick day" management regimen

Exclusion Criteria:

* Diagnosis of type 2 diabetes, or other types of diabetes (e.g. LADA).
* Treatment with an anti-hyperglycaemic agent (e.g., metformin, alpha-glucosidase inhibitors, pramlintide, glucagon-like peptide receptor agonist, etc.) within 3 months.
* Occurrence of severe hypoglycaemia involving coma/unconsciousness and/or seizure that required hospitalisation or hypoglycaemia-related treatment by an emergency physician or paramedic within 3 months.
* Hypoglycaemia unawareness based on Investigator judgement or frequent episodes of unexplained hypoglycaemia (2 or more unexplained episodes within 3 months).
* Occurrence of diabetic ketoacidosis within 6 months prior to study enrolment.
* Acute coronary syndrome (non-STEMI, STEMI and unstable angina pectoris), stroke or transient ischemic attack within 6 months.
* Any other clinical condition that, based on Investigator's judgement, would jeopardize patient safety during trial participation or would affect the study outcome (e.g., immunocompromised patients, patients who might be at higher risk of developing urinary, genital or mycotic infections, patients with chronic viral infections, etc.).
* Treatment with an SGLT2i within 30 days of Visit 1.
* NT-proBNP > 600 pg/mL
* Hemoglobin < 90 g/L
* Diagnosis of severe edema (per investigator judgment) within 3 months of screening
* Diagnosis of heart failure (NYHC stage III or IV).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Urine Albumin-Creatinine Ratio (UACR) | 4 weeks
  Primary: change from baseline in Urine Albumin-Creatinine Ratio (UACR) when treated with SC0062 alone versus combination of dapagliflozin and SC0062.

SECONDARY OUTCOMES:
Change from baseline in mGFR | 4 weeks
  Glomerular Filtration Rate (GFR) using iohexol clearance techniques.
Change in biomarkers of fluid retention | 4 weeks
  Change from baseline biomarkers of fluid retention (body weight, hemoglobin, N-terminal prohormone of Brain Natriuretic Peptide (NT-proBNP))
Change in biomarkers of fluid retention | 4 weeks
  Change from baseline biomarkers of fluid retention (Body Weight)
Change in biomarkers of fluid retention | 4 weeks
  Change from baseline biomarkers of fluid retention (hemoglobin)
Change in biomarkers of fluid retention | 4 weeks
  Change from baseline biomarkers of fluid retention (N-terminal prohormone of Brain Natriuretic Peptide (NT-proBNP))
Change from baseline Extracellular Volume (ECV) | 4 weeks
  Extracellular volume (ECV) using iohexol clearance techniques and bioimpedance spectroscopy.
Change from baseline blood pressure | 4 weeks
  Change in blood pressure as measure in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Hiddo J Lambers Heerspink, PhD, PharmD, Principal Investigator — University Medical Center Groningen
Locations (7):
- Denmark (3):
  - Steno Diabetes Center Aarhus, Aarhus
  - Steno Diabetes Center Copenhagen, Copenhagen
  - Regionshospitalet Gødstrup, Herning
- Finland (2):
  - University of Helsinki, Helsinki, Uusimaa
  - Turku University Hospital, Turku
- Netherlands (2):
  - Amsterdam University Academic Center, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen, Provincie Groningen

IPD SHARING:
Plan to Share IPD: No